CLINICAL TRIAL: NCT00918476
Title: A Phase 1, Open Label Fixed Sequence Study To Investigate The Effects Of Multiple Oral Doses Of Filibuvir On The Steady State Pharmacokinetics Of Oral Contraceptive Steroids In Healthy Female Subjects
Brief Title: Investigation Of The Effect Of Steady State Filibuvir On The Pharmacokinetics Of Oral Contraceptives (Levonorgestrel And Ethinyl Estradiol)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Model: Crossover | Masking: None
Other Study IDs: A8121008
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — filibuvir; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1. filibuvir + Oral Contraceptives (Experimental)
  Interventions: Drug: filibuvir + Oral Contraceptives

INTERVENTIONS:
Drug: filibuvir + Oral Contraceptives — This is an open-label, fixed sequence study to investigate the effect of filibuvir (600 mg BID on the pharmacokinetics of oral contraceptives steroids. Sixteen subjects who have been on any combination of ethinyl estradiol and levonorgesterol oral contraceptives for at least one consecutive month prior to Period 1 will be enrolled into the study. The study will be conducted over two 28 day menstrual cycles and Day 1 of each period is defined as the first day of dosing OC in each cycle. During the first cycle (Period 1), the subjects will receive OC QD for 21 days and filibuvir BID on Days 22 through 28. During the second cycle (Period 2) the subjects will receive OC QD and filibuvir BID for 21 days. The dosing of filibuvir will start in Period 1 (Days 22 - 28).

SUMMARY:
The purpose of this study is to estimate the effect of filibuvir on the pharmacokinetics of ethinyloestradiol [EE] and levonorgestrel [LN], to assess the safety and tolerability of 600 mg BID of filibuvir in healthy women and to investigate the pharmacokinetics of 600 mg BID of filibuvir in healthy women.

DETAILED DESCRIPTION:
To investigate the effects of multiple oral doses of filibuvir on the steady state pharmacokinetics of oral contraceptive steroids in healthy female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects between the ages of 18 and 45 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Subjects must have been on any combination of ethinyl estradiol and levonorgesterol oral contraceptives for at least one consecutive month prior to Period 1.
* Body Mass Index (BMI) of approximately 17.5 to 30.5 kg/m2; and a total body weight >45 kg.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
* Must be willing to practice an alternative method of contraception for the duration of the study in addition to oral contraceptive use.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any medical reason which would contraindicate the administration of oral contraceptives (as per label). Including but not limited to history of unexplained vaginal bleeding, current breast cancer, active liver disease, uncontrolled hypertension, history of diabetes with vascular complications, history of venous thrombosis, stroke, ischemic heart disease, history of severe headaches with focal neurologic symptoms.
* Female subjects of non-childbearing potential who meet the following criteria:
* Post menopausal, aged between 45-55 who have been amenorrheic for >2 years and who meet the criteria for serum FSH levels (>30 IU/L), or
* Females who have undergone a hysterectomy, or
* Females who have undergone tubal ligation, or
* Females who have undergone bilateral oophorectomy.
* History of discontinued use of oral contraceptives for medical reasons.
* History of febrile illness within 5 days prior to the first dose.
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
AUCtau, Cmax, for LN and EE on Day 21 in Period 1 and Period 2. | 21 days

SECONDARY OUTCOMES:
LN and EE - Tmax and t1/2 (if data permit) in Period 1 and Period 2. Filibuvir - AUCtau, Cmax, Cmin, and Tmax on Day 28 of Period 1 and Day 21 of Period 2. | 21 days
Safety (AE, lab, vital, ECG, etc). | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8121008&StudyName=Investigation%20Of%20The%20Effect%20Of%20Steady%20State%20Filibuvir%20On%20The%20Pharmacokinetics%20Of%20Oral%20Contraceptives%20%28Levonorgestrel%20And%20Ethinyl%20Estradiol